CLINICAL TRIAL: NCT06909370
Title: The Effect of Peer Education for Human Papilloma Virus (HPV) on Knowledge, Awareness and Concern Levels of Students in the Faculty of Health Sciences
Brief Title: Peer Education on HPV: Impact on Health Sciences Students' Knowledge, Awareness, and Concern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Beyzanur İşbay Aydemir, Lecturer, Istanbul Aydın University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024/04
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Human Papilloma Virus (HPV)
Keywords: HPV; peer education; awareness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Hygiene Training (Experimental)
  Interventions: Behavioral: peer education

INTERVENTIONS:
Behavioral: peer education — The training titled "The Effect of Peer Education on Human Papillomavirus (HPV) for Students in the Faculty of Health Sciences on Knowledge, Awareness, and Concern Levels" includes scientific and up-to-date information about HPV transmission methods, prevention, risk factors, treatment methods, and vaccination. The content of the training aims to provide students with accurate information about HPV, as well as highlight the negative health effects of the virus, particularly its association with serious diseases like cervical cancer. The training seeks to increase students' awareness of HPV and help them manage their levels of concern about the virus. Through the peer education method, students were able to interact with each other, thus providing a more effective learning experience.

SUMMARY:
According to the World Health Organization (WHO), 400 million treatable sexually transmitted diseases (STDs) such as syphilis, chlamydia and human papillomavirus (HPV) occur each year in people aged 15-49, mostly in developing countries. As HPV is a sexually transmitted virus, it has been shown to be the most important aetiological factor in cervical cancer in women (99.7%). Vaccination and education of young people about sexuality and STDs are very important in the prevention of HPV. In this respect, the aim of this study was to find out the level of knowledge, concern and awareness of HPV infection among university students and to increase their awareness by informing them about the subject through their peers. The study was conducted as a pre-test and post-test one-group study. The sample of the study consisted of all final year students of Physiotherapy and Rehabilitation (85 students), Nutrition and Dietetics (60 students), Audiology (35 students), Child Development (80 students), Health Management (44 students) and Social Work (45 students) studying in the spring semester of the 2023-2024 academic year. The students were trained by the Gynaecology Nursing Intern student group (9 students) of the Department of Nursing. Data were collected using the Sociodemographic Characteristics Form, the HPV Knowledge Scale and the Human Papilloma Virus Awareness and Concern Level Scale (HPV-FAS). The relevant forms and the consent form were completed by the students before, after and one month after the training.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who are senior students in the Faculty of Health Sciences departments and who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Individuals who did not complete the study and did not speak and understand Turkish were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Characteristics Form | Through study completion, an average of 6 months
  It consists of nine questions containing sociodemographic data of students, developed by the researchers.
HPV Knowledge Scale (HPV-KS) | Through study completion, an average of 6 months
  The HPV-KS was developed in 2013 by Waller and colleagues to measure individuals' knowledge levels about HPV, the HPV vaccine, and screening tests. The scale examines whether individuals have previously heard about HPV, the HPV vaccine, and HPV screening tests, as well as the extent of their knowledge on these topics. The first subdimension of the HPV-KS consists of 16 items and assesses participants' general knowledge about HPV. The second subdimension includes six items and is related to HPV screening tests. The third subdimension consists of seven items and asks participants to respond to items about the HPV vaccine. The independent subdimension of the HPV-KS has been developed in three different forms for the HPV vaccination program conducted in three different countries. For each item in the HPV-KS, participants are expected to mark "Yes," "No," or "I don't know." The total score obtained from the HPV-KS ranges from 0 to 33.
Human Papillomavirus Awareness and Concern Scale (HPV-ACS) | Through study completion, an average of 6 months
  Developed by Yılmaz Esencan and colleagues (2023), this scale is designed as a five-point Likert-type and consists of 19 items and three subdimensions. The subdimensions of the scale are "Concern about health," "Concern about being excluded," and "Awareness." The scale scores range from a minimum of 0 to a maximum of 76 points. A higher total score indicates a stronger awareness of HPV. The Cronbach's Alpha reliability coefficient of the original scale was determined to be 0.905.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided